CLINICAL TRIAL: NCT02253134
Title: Monitoring of Syncopes and/or Sustained Palpitations of Suspected Arrhythmic Origin With External Loop-Recorder (SpiderFLASH)
Acronym: ITHO04
Status: Completed | Type: Observational
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: SYNARR-FLASH STUDY - ITHO04
Record Dates: First submitted 2013-07-10; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Syncope; Palpitations
Keywords: Syncopal events; Palpitation events
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the diagnostic yield (at 1 month post enrollment) of an external loop recorder (SpiderFlash-T) in patients with syncope or palpitations of suspected arrhythmic origin, within 30 days before enrollment.

DETAILED DESCRIPTION:
Diagnostic yield (primary outcome) definition = Number of patients with conclusive diagnosis (as per investigators' decision) over the total number of patients

ELIGIBILITY:
Inclusion Criteria:

* Syncope and/or palpitations events occurred in the last 30 days
* Events likely of arrhythmic origin
* No conclusive diagnosis established yet
* High probability of episodes recurrence (presence of at least one previous event in the last 12 months)
* Patient has signed the consent to participate to the study and/or to data treatment

Exclusion Criteria:

* Inability to understand the purpose of the study or refusal to cooperate
* Expected low compliance with the recording technique.
* Logistical impossibility to deliver the ELR within 30 days after the index event (or after discharge from ER and/or hospitalization and/or clinic visit)
* Already included in other competitor clinical study
* Under guardianship
* Age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that present unexplained Syncope and/or palpitations events of a suspected arrhythmic origin
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2010-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the mean value of the diagnostic yield in one month | 1 month
  number of pts with a conclusive diagnosis (per investigators' decision) over the total number of patients

SECONDARY OUTCOMES:
Diagnostic yield of the ELR stratified by each kind of diagnosed event, by week and by event occurred post enrollment | 1 month
Recurrence rate stratified by syncope /palpitation, by week and by type of events occurred post enrollment | 1 month
Analysis of arrhythmic vs non arrhythmic findings stratified by kind of index events (syncope /palpitations) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela T Locati, Principal Investigator — Azienda Ospedaliera Niguarda Ca' Granda - Milano
Locations (10):
- UZ Gasthuisberg Leuven, Leuven, Belgium
- Italy (2):
  - Az. Sanit. Locale N. 4 Chiavarese, Lavagna
  - Ospedale Niguarda Ca Granda, Milan
- Hospital de Santa Marta, Lisbon, Portugal
- Spain (5):
  - Institut Universitari Dexeus, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario 12 de Octubre, Madrid
- Universitätsklinik für Kardiologie Inselspital, Bern, Switzerland